CLINICAL TRIAL: NCT03736018
Title: A Randomised Controlled Trial Assessing the Value of Computed Tomography Cardiac Angiography in Improving Patient Satisfaction and Reducing Contrast Load, Procedural Duration and Complications in Patients Who Had Previous Bypass Operation Undergoing Invasive Coronary Angiography
Brief Title: Randomised Controlled Trial to Assess Whether Computed Tomography Cardiac Angiography Can Improve Invasive Coronary Angiography in Bypass Surgery Patients
Acronym: BYPASS-CTCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Reda 012466
Record Dates: First submitted 2018-11-05; First posted 2018-11-08 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Ischaemic Heart Disease; Contrast-induced Nephropathy
Keywords: Coronary Artery Bypass Grafts; Computed Tomography Cardiac Angiography; Invasive Coronary Angiogram
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTCA + ICA (Active Comparator): Computed Tomography Cardiac Angiography (CTCA) performed prior to invasive coronary angiogram (ICA).
  Interventions: Diagnostic Test: CTCA
- ICA only (No Intervention): Invasive coronary angiogram (ICA) performed only.

INTERVENTIONS:
Diagnostic Test: CTCA — Computed Tomography Cardiac angiography (CTCA) performed prior to invasive coronary angiogram (ICA).
  Other Names: Computed Tomography Cardiac angiography
  Arms: CTCA + ICA

SUMMARY:
A large number of patients with symptomatic ischaemic heart disease undergo coronary artery bypass grafting (CABG) to alleviate their symptoms and improve prognosis. Given the progressive nature of coronary disease, bypass grafts can narrow or block over time, leading to chest pain and the need for further invasive coronary angiography. Invasive coronary procedures in patients with bypass grafts can be more complicated due to the variation in bypass graft ostia. This can lead to longer procedure times, with higher doses of contrast and radiation and more discomfort for the patient. The aim of this study is to see if the use of computed tomography cardiac angiography (CTCA) in patients with previous bypass grafts prior to invasive coronary angiography will help make their procedure safer and quicker.

DETAILED DESCRIPTION:
The BYPASS-CTCA trial is a single-centre, randomised controlled trial, which plans to recruit 688 patients who have had previous bypass grafts and require invasive coronary angiography over a period of 30 months.

Patients will be randomised to receive either computed tomography cardiac angiography (CTCA) prior to their invasive coronary angiogram, or invasive coronary angiography alone.

The primary endpoints will be the incidence of contrast induced nephropathy, the duration of the invasive coronary angiographic procedure and patient satisfaction. A number of secondary endpoints will also be looked at.

Findings from BYPASS-CTCA will potentially demonstrate that a CTCA prior to invasive coronary angiography in this cohort of patients reduces the incidence of contrast-induced kidney injury, the length of procedure and improves patients satisfaction. The results of this trial may influence future clinical practice guidelines in coronary artery bypass graft patients undergoing invasive coronary procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing invasive coronary angiogram +/- percutaneous coronary Intervention
2. Previous Coronary Artery Bypass Grafting (CABG)
3. Aged ≥18
4. Patients able and willing to give their written informed consent.

Exclusion Criteria:

1. Subjects presenting with ST elevation myocardial infarction, cardiogenic shock (systolic blood pressure <80 mmHg for >30 minutes, or requiring inotropes or emergency intra aortic balloon pump for hypotension treatment) or cardiopulmonary resuscitation.
2. Subjects with eGFR <20ml/min or on renal replacement therapy.
3. Current life-threatening condition other than vascular disease that may prevent a subject completing the study.
4. Clinical instability including cardiogenic shock, hypotension (low blood pressure-systolic blood pressure less than 90 mmHg), sustained ventricular or atrial arrhythmia requiring intravenous medications.
5. Inability to tolerate beta-blockers, including those with chronic obstructive pulmonary disease or asthma, complete heart block, second-degree atrioventricular block
6. Known contrast dye allergy.
7. Pregnancy or unknown pregnancy status.
8. Patients considered unsuitable to participate by the research team (e.g., due to medical reasons, laboratory abnormalities, or subject's unwillingness to comply with all study related procedures).
9. Inability or refusal to provide informed consent.
10. Any inclusion criteria not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Procedural duration | Interval between administration of local anaesthesia for obtaining vascular access and removal of the last catheter
  Length of invasive coronary angiogram
Incidence of Contrast Induced Nephropathy | 48-72hours
  Defined by Kidney Disease: Improving Global outcomes (KDIGO) criteria
Patient satisfaction | 4-6hours
  Patient satisfaction measured by validated questionnaire

SECONDARY OUTCOMES:
Contrast amount | From time of arterial sheath insertion to removal of arterial catheters
  Contrast amount (mls) administered during invasive coronary angiogram
Radiation exposure | From time of arterial sheath insertion to removal of arterial catheters
  Radiation exposure (mSv) during invasive coronary angiogram
Angiography related complications | 4-6hours
  Angiography related complications (coronary or aortic dissection, stroke, bleeding, vascular access complications)
Radial access rate | From time of randomisation to end of invasive coronary angiogram procedure
  Radial access rates during invasive coronary angiogram
Catheters used | From time of arterial sheath insertion to removal of arterial catheters
  Number of catheters used during invasive coronary angiogram
Computed Tomography Cardiac Angiography accuracy | From time of randomisation to end of invasive coronary angiogram procedure
  Accuracy of the Computed Tomography Cardiac Angiography scan for detecting graft patency
Number of grafts not identified | From time of arterial sheath insertion to removal of arterial catheters
  Number of grafts not identified during invasive coronary angiogram
Cost effectiveness of computed tomography cardiac angiography | 12 months
  Incremental Cost Effectiveness Ratio (ICER)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Jones, MRCP, PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Trial protocol to be published
Supporting Information: Study Protocol
Time Frame: Late 2018
Access Criteria: Freely available via journal

REFERENCES:
- [Derived] Kelham M, Beirne AM, Rathod KS, Andiapen M, Wynne L, Learoyd AE, Forooghi N, Ramaseshan R, Moon JC, Davies C, Bourantas CV, Baumbach A, Manisty C, Wragg A, Ahluwalia A, Pugliese F, Mathur A, Jones DA. CTCA Prior to Invasive Coronary Angiography in Patients With Previous Bypass Surgery: Patient-Related Outcomes, Imaging Resource Utilization, and Cardiac Events at 3 Years From the BYPASS-CTCA Trial. Circ Cardiovasc Interv. 2024 Dec;17(12):e014142. doi: 10.1161/CIRCINTERVENTIONS.124.014142. Epub 2024 Nov 25. PMID 39584261
- [Derived] Kelham M, Beirne AM, Rathod KS, Andiapen M, Wynne L, Ramaseshan R, Learoyd AE, Forooghi N, Moon JC, Davies C, Bourantas CV, Baumbach A, Manisty C, Wragg A, Ahluwalia A, Pugliese F, Mathur A, Jones DA; BYPASS-CTCA Trial Investigators. The effect of CTCA guided selective invasive graft assessment on coronary angiographic parameters and outcomes: Insights from the BYPASS-CTCA trial. J Cardiovasc Comput Tomogr. 2024 May-Jun;18(3):291-296. doi: 10.1016/j.jcct.2024.03.004. Epub 2024 Mar 11. PMID 38462389
- [Derived] Jones DA, Beirne AM, Kelham M, Rathod KS, Andiapen M, Wynne L, Godec T, Forooghi N, Ramaseshan R, Moon JC, Davies C, Bourantas CV, Baumbach A, Manisty C, Wragg A, Ahluwalia A, Pugliese F, Mathur A; BYPASS-CTCA Trial Committees and Investigators. Computed Tomography Cardiac Angiography Before Invasive Coronary Angiography in Patients With Previous Bypass Surgery: The BYPASS-CTCA Trial. Circulation. 2023 Oct 31;148(18):1371-1380. doi: 10.1161/CIRCULATIONAHA.123.064465. Epub 2023 Sep 29. PMID 37772419
- [Derived] Beirne AM, Rathod KS, Castle E, Andiapen M, Richards A, Bellin A, Hammond V, Godec T, Moon JC, Davies C, Bourantas CV, Wragg A, Ahluwalia A, Pugliese F, Mathur A, Jones DA. The BYPASS-CTCA Study: the value of Computed Tomography Cardiac Angiography (CTCA) in improving patient-related outcomes in patients with previous bypass operation undergoing invasive coronary angiography: Study Protocol of a Randomised Controlled Trial. Ann Transl Med. 2021 Sep;9(17):1395. doi: 10.21037/atm-21-1455. PMID 34733947